CLINICAL TRIAL: NCT00379067
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Effect of Tamsulosin OCAS 0.4 mg Tablets, Once Daily on Nocturia, Compared to Placebo, in Patients With Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia
Brief Title: A Phase 4 Study With Tamsulosin OCAS to Assess Nighttime Voiding.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe Ltd. (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 617-EC-006
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Nocturia; Actigraphy; Tamsulosin
MeSH Terms: conditions — Prostatic Hyperplasia; Nocturia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Tamsulosin OCAS tablet
  Interventions: Drug: Tamsulosin OCAS
- 2 (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin OCAS — Adrenoceptor antagonist
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
Randomized, double-blind, placebo-controlled study with two treatment arms (Tamsulosin OCAS 0.4 mg & placebo). The study comprises a 2-week placebo run-in followed by a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having LUTS associated with BPH
* On average, at least 2 voids per night over the last week
* A maximum of 4 hours of undisturbed sleep expected per night (night time is defined as the time from going to bed with the purpose of sleeping until waking up with the purpose of getting up)

Exclusion Criteria:

* Subject is currently taking diuretics
* Subjects who work shift hours and whose hours of work include any time between 23.00 and 06.00h

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2005-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The change from baseline to week 12 in mean number of nocturnal voids | 12 weeks

SECONDARY OUTCOMES:
The change from baseline to week 12 in mean hours of undisturbed sleep, defined as the time from falling asleep to first awakening to void | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Medical Affairs Europe, Astellas Pharma Europe Limited, Lovett House, Lovett Road, Staines Middlesex TW 18 3AZ